CLINICAL TRIAL: NCT06335199
Title: Movement-Associated tVNS and Responsiveness Testing for Personalized Rehabilitation
Brief Title: tVNS Responsiveness Testing With Pupil Size
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Georgia Institute of Technology (Other)
Collaborators: Emory University (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Basic Science
Other Study IDs: H24109; 5P2CHD086844-09 (NIH)
Record Dates: First submitted 2024-03-15; First posted 2024-03-28 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-03

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Unilateral Left tVNS (Experimental): Electrical stimulation to the vagus nerve area of the outer ear on the left side.
  Interventions: Procedure: Unilateral Left tVNS stimulation
- Bilateral tVNS (Experimental): Electrical stimulation to the vagus nerve area of the outer ear on both sides.
  Interventions: Procedure: Bilateral tVNS stimulation
- Unilateral Left Sham (Sham Comparator): Electrical stimulation to the non-vagus nerve area of the outer ear on the left side.
  Interventions: Procedure: Unilateral Left Sham stimulation
- Bilateral Sham (Sham Comparator): Electrical stimulation to the non-vagus nerve area of the outer ear on both sides.
  Interventions: Procedure: Bilateral Sham stimulation
- Unilateral Right tVNS (Experimental): Electrical stimulation to the vagus nerve area of the outer ear on the right side.
  Interventions: Procedure: Unilateral Right tVNS stimulation
- Unilateral Right Sham (Sham Comparator): Electrical stimulation to the non-vagus nerve area of the outer ear on the right side.
  Interventions: Procedure: Unilateral Right Sham stimulation

INTERVENTIONS:
Procedure: Unilateral Left tVNS stimulation — Electrical stimulation to the cymba concha or tragus (depending on the ear dimension) of the outer ear on the left side after successful trials.
  Arms: Unilateral Left tVNS
Procedure: Bilateral tVNS stimulation — Electrical stimulation to the cymba concha or tragus (depending on the ear dimension) of the outer ear on both sides after successful trials.
  Arms: Bilateral tVNS
Procedure: Unilateral Left Sham stimulation — Electrical stimulation to the earlobe of the outer ear on the left side after successful trials.
  Arms: Unilateral Left Sham
Procedure: Bilateral Sham stimulation — Electrical stimulation to the earlobe of the outer ear on both sides after successful trials.
  Arms: Bilateral Sham
Procedure: Unilateral Right tVNS stimulation — Electrical stimulation to the cymba concha or tragus (depending on the ear dimension) of the outer ear on the right side after successful trials.
  Arms: Unilateral Right tVNS
Procedure: Unilateral Right Sham stimulation — Electrical stimulation to the earlobe of the outer ear on the right side after successful trials.
  Arms: Unilateral Right Sham

SUMMARY:
The goal of this study is to learn about the acute pupil response to transcutaneous vagus nerve stimulation (tVNS) in stroke survivors and healthy adults. The main question it aims to answer is whether pupil size response is greater with bilateral tVNS compared to unilateral tVNS. Participants will receive tVNS and sham at the outer ear unilaterally and bilaterally in resting condition. The pupil size of the participants will be recorded during tVNS.

DETAILED DESCRIPTION:
Participants will wear surface electrodes on the outer ear on both sides and a finger device that monitors heart rate. The attachment sites are the tragus or the cymba concha (depending on the shape and size of the ear) for tVNS and the ear lobe for sham. The electrical current will have a pulse duration of 0.1 ms at 30 Hz with an intensity below the pain threshold or 5 milliamp, whichever is lower, for a duration of 0.5 s. The experimental stimulation intensity will be determined as just below the pain threshold. Participants will receive multiple blocks of unilateral and bilateral stimulations to the sham or tVNS electrodes at rest, during which their pupil size will be recorded. The order of unilateral/bilateral and sham/tVNS stimulation will be randomized.

ELIGIBILITY:
Inclusion Criteria:

* 18-89 years old across all races, genders, and ethnicities.
* Post-stroke subjects will have persistent hemiparesis on the upper extremity (UE) with some residual UE voluntary movement.

Exclusion Criteria:

Able-bodied subjects:

* Younger than 18 years old or older than 89 years old
* Current or history of cardiac disease
* Have a vision problem not corrected by glasses or contact lenses
* Have an implanted device such as a neurostimulator or cochlear implant
* Current or history of tympanic membrane perforation
* Had a stroke or lesion (including tumor) in your brain
* Had a head injury or brain surgery
* Suffer from frequent or severe headaches
* Had a fainting spell or syncope
* Have any metal in the head such as shrapnel, surgical clips, or fragments from welding or metal work
* Have any implanted device such as cardiac pacemakers, medical pumps, or intra-cardiac lines
* Had any brain-related conditions (i.e. multiple sclerosis, Parkinson, Alzheimer)
* Had any illness that caused brain injury (i.e. meningitis, aneurysm, brain tumor)
* Had any head trauma that was associated with a loss of consciousness or diagnosed as a concussion
* Being treated for any psychiatric condition (i.e. depression, anxiety, PTSD, schizophrenia)
* Suspected of pregnancy

Post-stroke subjects:

* Younger than 18 years old or older than 89 years old
* Current or history of cardiac disease
* Have a vision problem not corrected by glasses or contact lenses
* Have any implanted devices such as a neurostimulator or cochlear implant
* Current or history of tympanic membrane perforation
* No persistent hemiparesis on the upper extremity (UE)
* No residual UE voluntary movement
* A first stroke less than 4 months prior to the participation
* Serious uncontrolled medical conditions
* Excessive pain in any joint of the more affected extremity
* Unable to stand independently for 2 min., transfer independently to and from the toilet or perform sit-to-stand
* Suffer from frequent or severe headaches
* Had a fainting spell or syncope
* Have any metal in the head such as shrapnel, surgical clips, or fragments from welding or metal work
* Have any implanted device such as cardiac pacemakers, medical pumps, or intra-cardiac lines
* Had any illness that caused brain injury (i.e. meningitis, aneurysm, brain tumor)
* Had any head trauma that was associated with a loss of consciousness or diagnosed as a concussion
* Being treated for any psychiatric condition (i.e. depression, anxiety, PTSD, schizophrenia)
* Suspected of pregnancy
* A score of less than 24 on the Folstein Mini-Mental State Examination
* Excessive frailty or lack of stamina (e.g., cannot attend to instructions, stay awake, engage in functional activities, etc.)
* Excessive pain in any joint of the more affected extremity that could limit ability to cooperate with the intervention

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2024-11-14 (Actual); Primary Completion 2025-10-27 (Actual); Study Completion 2025-10-27 (Actual)

PRIMARY OUTCOMES:
Pupil size change | Day 1
  Acute change in pupil size in response to electrical stimulation, relatively expressed as a percent change from the baseline

CONTACTS AND LOCATIONS:
Overall Officials: Minoru Shinohara, Ph.D., Principal Investigator — Georgia Institute of Technology
Locations (1):
- Human Neuromuscular Physiology Lab, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data on pupil size change will be available to other researchers outside the primary research group.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data will become available after the publication of all papers from the study.
Access Criteria: The scientific data will be made available by a data repository after approval.

DOCUMENTS (1):
  • Informed Consent Form (2025-08-06): https://cdn.clinicaltrials.gov/large-docs/99/NCT06335199/ICF_000.pdf